CLINICAL TRIAL: NCT06813989
Title: Evaluation of the Effectiveness of Carotid Flow Measurements in Predicting Post-Spinal Hypotension in Pregnant Women
Brief Title: Carotid Flow Measurements in Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2025
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Postspinal Hypotension; Pregnant Women Undergoing Cesarean Delivery
Keywords: carotid blood flow; corrected carotid flow time; postspinal hypotension; cesarean delivery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postspinal hypotension: Hypotension will be defined as (1) a decrease in systolic blood pressure >30% or a decrease in mean arterial pressure (MAP) >20% from baseline, or (2) systolic blood pressure <90 mmHg or MAP <65 mmHg, within the time period starting from spinal anaesthesia and surgical delivery.
  Interventions: Other: carotid ultrasound

INTERVENTIONS:
Other: carotid ultrasound — The investigator will perform a carotid ultrasound just 2 cm before the carotid bulb and measure the corrected flow time and flow using Doppler and pulse wave analysis. The corrected carotid flow time will be calculated according to Bazett's equation.

SUMMARY:
The goal of this observational study is to reveal the relation between carotid flow changes and post-spinal hypotension in pregnant women between the ages of 20-40. The main question it aims to answer is:

Do the carotid flow blood flow measurements and corrected flow time change before and after spinal anaesthesia related to postspinal hypotension? Participants are already receiving spinal anaesthesia to receive a caesarean section. As part of their regular anaesthesia management protocol, they will answer questions about anaesthesia management. The participants will only examined by ultrasound twice.

DETAILED DESCRIPTION:
In this study, Doppler ultrasound measurements will be taken to evaluate the diameter and flow velocity of the left carotid artery in pregnant women aged 20-40 years, classified as ASA 1-2 term and uncomplicated, upon their arrival at the operating room in the supine position. Measurements will be performed three times at the cricoid level, before the carotid bifurcation, and directly from the arch to mitigate any errors due to the measurer. These measurements will be conducted by the same individual (B.C) and repeated three minutes after returning to the supine position post-spinal anaesthesia, with changes between the two measurements recorded.

The spinal anaesthesia dose will be standardized with 10 mg of heavy bupivacaine and 10 mcg of fentanyl. Hemodynamic data from the time patients enter the operating room until baby delivery will be recorded.

Hypotension during this period will be defined as (1) a decrease in systolic blood pressure >30% or a decrease in mean arterial pressure (MAP) >20% from baseline, or (2) systolic blood pressure <90 mmHg or MAP <65 mmHg. Carotid flow measurements and the amount of crystalloid administered during spinal anaesthesia will be noted in hypotensive and non-hypotensive patients.

ELIGIBILITY:
Inclusion Criteria:

* "Uncomplicated term pregnant women aged 20-40 years classified as ASA 1-2.

Exclusion Criteria:

* Those diagnosed with preeclampsia or eclampsia or with systolic blood pressure above 160

Individuals with arrhythmia

Individuals with contraindications for spinal anesthesia

Individuals with Ba MI over 40

Those with a gestational age under 36 weeks or over 41 weeks

Individuals with chronic kidney insufficiency (GRF under 60)

Those with carotid stenosis or a history of previous cerebrovascular events

Patients with placental anomalies

Those initially planned for expected delivery but later switched to cesarean after being taken to trauma.

Patients were taken to the operating room with an emergency cesarean decision

In case of failed spinal anaesthesia, those who switched to general anaesthesia before delivery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women scheduled for cesarean section
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
postspinal hypotension | from spinal anaesthesia till surgical delivery
  Hypotension is defined as (1) a decrease in systolic blood pressure >30% or a decrease in mean arterial pressure (MAP) >20% from baseline, or (2) systolic blood pressure <90 mmHg or MAP <65 mmHg.

SECONDARY OUTCOMES:
fluid resuscitation | from spinal anaesthesia till surgical delivery
  amount of fluid given for co loading during anaesthesia application

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim HJ, Cho AR, Lee H, Kim H, Kwon JY, Lee HJ, Kang C, Jeon S, Kim N. Ultrasonographic Carotid Artery Flow Measurements as Predictors of Spinal Anesthesia-Induced Hypotension in Elderly Patients: A Prospective Observational Study. Med Sci Monit. 2022 Nov 28;28:e938714. doi: 10.12659/MSM.938714. PMID 36437555
- [Result] Kim HJ, Choi YS, Kim SH, Lee W, Kwon JY, Kim DH. Predictability of preoperative carotid artery-corrected flow time for hypotension after spinal anaesthesia in patients undergoing caesarean section: A prospective observational study. Eur J Anaesthesiol. 2021 Apr 1;38(4):394-401. doi: 10.1097/EJA.0000000000001376. PMID 33122575